CLINICAL TRIAL: NCT06641843
Title: Magnetic Resonance Myocardial Stress Perfusion: to Improve the Myocardial Evaluation in Pediatric Patients with Cardiovascular Disease
Brief Title: Magnetic Resonance Myocardial Stress Perfusion in Pediatric Patients with Cardiovascular Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ling-Yi Wen, Principal Investigator, West China Second University Hospital
Other Study IDs: WestChinaSUH2024223
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Kawasaki Disease; Cardiovascular Disease; Anomalous Origin of Coronary Artery
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The whole boold including blood cell and plasma will be collected for laboratory test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosed with cardiovascular disease: Patients diagnosed with cardiovascular disease, including Kawasaki disease, anomalous origin of coronary artery, postoperative congenital heart diseases

SUMMARY:
the goal of this observational study is to evaluate myocardial ischemia and myocardial microcirculation dysfunction in children with cardiovascular disease by myocardial stress perfusion imaging.

During their disease progress, participants will undergo myocardial stress perfusion, laboratory tests when hospitalization and follow-up, and the baseline data will be collected in the admission. all the above examination data will be analysed to identify early subclinical myocardial changes and evaluate the value of magnetic resonance myocardial stress perfusion in predicting prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cardiovascular disease, including Kawasaki disease, anomalous origin of coronary artery, postoperative congenital heart disease.

Exclusion Criteria:

* Mental abnormalities or poor compliance ; heart, kidney and other important organs were seriously incomplete.
* MRI examination contraindications ; gadolinium contrast agent contraindications ; claustrophobia.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From September 2024 to Jaunary 2034, pediatric patients diagnosed with cardiovascular disease were prospectively recruited from West China Second University Hospital, Sichuan University.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2034-09-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovscualr events | 10 years after the onset
  Major adverse cardiovascular events including cardiac death, transient ischemic attack or stroke, myocardial infarction, arrhythmia, heart failure, severe valvular disease, percutaneous coronary intervention, coronary artery bypass graft, and other cardiovascular surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University., Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou W, Lee JCY, Leung ST, Lai A, Lee TF, Chiang JB, Cheng YW, Chan HL, Yiu KH, Goh VK, Pennell DJ, Ng MY. Long-Term Prognosis of Patients With Coronary Microvascular Disease Using Stress Perfusion Cardiac Magnetic Resonance. JACC Cardiovasc Imaging. 2021 Mar;14(3):602-611. doi: 10.1016/j.jcmg.2020.09.034. Epub 2020 Nov 25. PMID 33248966
- [Background] Erbel C, Mukhammadaminova N, Gleissner CA, Osman NF, Hofmann NP, Steuer C, Akhavanpoor M, Wangler S, Celik S, Doesch AO, Voss A, Buss SJ, Schnabel PA, Katus HA, Korosoglou G. Myocardial Perfusion Reserve and Strain-Encoded CMR for Evaluation of Cardiac Allograft Microvasculopathy. JACC Cardiovasc Imaging. 2016 Mar;9(3):255-66. doi: 10.1016/j.jcmg.2015.10.012. PMID 26965729
- [Background] Shaw JL, Nelson MD, Wei J, Motwani M, Landes S, Mehta PK, Thomson LEJ, Berman DS, Li D, Bairey Merz CN, Sharif B. Inverse association of MRI-derived native myocardial T1 and perfusion reserve index in women with evidence of ischemia and no obstructive CAD: A pilot study. Int J Cardiol. 2018 Nov 1;270:48-53. doi: 10.1016/j.ijcard.2018.06.086. Epub 2018 Jun 22. PMID 30041981
- [Background] Park SM, Wei J, Cook-Wiens G, Nelson MD, Thomson L, Berman D, Handberg E, Petersen J, Anderson D, Pepine CJ, Merz CNB. Left ventricular concentric remodelling and functional impairment in women with ischaemia with no obstructive coronary artery disease and intermediate coronary flow reserve: a report from the WISE-CVD study. Eur Heart J Cardiovasc Imaging. 2019 Aug 1;20(8):875-882. doi: 10.1093/ehjci/jez044. PMID 30904924
- [Background] Gulati M, Levy PD, Mukherjee D, Amsterdam E, Bhatt DL, Birtcher KK, Blankstein R, Boyd J, Bullock-Palmer RP, Conejo T, Diercks DB, Gentile F, Greenwood JP, Hess EP, Hollenberg SM, Jaber WA, Jneid H, Joglar JA, Morrow DA, O'Connor RE, Ross MA, Shaw LJ. 2021 AHA/ACC/ASE/CHEST/SAEM/SCCT/SCMR Guideline for the Evaluation and Diagnosis of Chest Pain: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Nov 30;144(22):e368-e454. doi: 10.1161/CIR.0000000000001030. Epub 2021 Oct 28. PMID 34709928
- [Background] Ferrari R, Rosano G. 2019 guidelines for the diagnosis and management of chronic coronary syndromes: congratulations and criticism. Eur Heart J Cardiovasc Pharmacother. 2020 Sep 1;6(5):331-332. doi: 10.1093/ehjcvp/pvaa006. No abstract available. PMID 32154890
- [Background] Aetesam-Ur-Rahman M, Brown AJ, Jaworski C, Giblett JP, Zhao TX, Braganza DM, Clarke SC, Agrawal BSK, Bennett MR, West NEJ, Hoole SP. Adenosine-Induced Coronary Steal Is Observed in Patients Presenting With ST-Segment-Elevation Myocardial Infarction. J Am Heart Assoc. 2021 Jul 6;10(13):e019899. doi: 10.1161/JAHA.120.019899. Epub 2021 Jun 30. PMID 34187187
- [Background] Patel AR, Salerno M, Kwong RY, Singh A, Heydari B, Kramer CM. Stress Cardiac Magnetic Resonance Myocardial Perfusion Imaging: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Oct 19;78(16):1655-1668. doi: 10.1016/j.jacc.2021.08.022. PMID 34649703